CLINICAL TRIAL: NCT01045746
Title: Effects of Stochastic Resonance Therapy on Postural Control in the Elderly Population (Pilot Study)
Brief Title: Effects of Whole-Body Vibration on Balance in the Elderly Population
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bern University of Applied Sciences (Other)
Collaborators: Swiss Federal Institute of Technology (Other); Maastricht University Medical Center (Other); Goethe University (Other)
Responsible Party: Principal Investigator, Slavko Rogan, cand. PhD, PTMsc, MSc PT, Bern University of Applied Sciences
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: PhD pilot study I
Record Dates: First submitted 2010-01-08; First posted 2010-01-11 (Estimated); Last update posted 2014-12-23 (Estimated); Status verified 2014-12

CONDITIONS: Distorted; Balance
Keywords: whole-body vibration; stochastic resonance Therapy; static balance; balance, mobility; elderly, reaction time; The focus of the study is effect of SRT on postural balance

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group 1 (Experimental): T0, Stochastic resonance whole-body vibration A intervention over four weeks, three time a week;T1, 16 days wash-out period; T2, Stochastic resonance whole-body vibration B intervention over four weeks, three times week, T3
  Interventions: Device: Stochastic resonance whole-body vibration A; Device: Stochastic resonance whole-body vibration b
- Group 2 (Experimental): T0, Stochastic resonance whole-body vibration B intervention over four weeks, three time a week;T1, 16 days wash-out period;T2, Stochastic resonance whole-body vibration A intervention over four weeks, three times week, T3
  Interventions: Device: Stochastic resonance whole-body vibration A; Device: Stochastic resonance whole-body vibration b

INTERVENTIONS:
Device: Stochastic resonance whole-body vibration A — over four weeks, three times a week with 5 Hz, Noise 4 and than over four weeks three times a week with 1 Hz, Noise 1.
  Other Names: Zeptor med ®
Device: Stochastic resonance whole-body vibration b — over four weeks, three times a week with 1 Hz, Noise 1 and than four weeks three times a week with 5 Hz, Noise 4.
  Other Names: Zeptor med ®

SUMMARY:
The goal of this pilot study is to test whether in the elderly population there are acute long-term improvements in both the static and dynamic balance, reaction time and mobility with the use of WBV.

DETAILED DESCRIPTION:
Exercise therapy plays an important role in health promotion, preservation of physical function and in preventing loss of independence among the elderly. They work beside an improvement in balance, a positive effect on metabolic and cardiovascular disorders, reducing falls, osteoporosis, colon cancer, breast cancer, depression, anxiety, and the general well-being. There is preliminary evidence to indicated that balance, and strength can be trained in the elderly using whole-body vibration (WBV) therapy. The use of WBV in the elderly population has shown to be a simple and effective treatment in the areas of balance and mobility. It would be very desirable to investigate these factors further in order to provide evidence for the delivery of sustainability of training methods.

ELIGIBILITY:
Inclusion Criteria:

* BESA to include performance level 0,1,2.
* live in the senior residence Multengut Muri or in the canton of Bern.
* apart from the complaints of old age healthy and can stand with or without aids.
* more than 22 points at the Mini-Mental State Examination

Exclusion Criteria:

* Seniors / graduates may no severe, uncorrected visual disturbances (eg, low vision, double vision, skew deviation).
* Acute stress the incompatibility of the lower limb / hip / ridge during the SRT: joint disease, thrombosis, fresh fractures, infections, tissue damage, or fresh surgical scars.
* Seniors / inside with lower leg-/thigh prostheses.
* alcoholics.

Ages: 65 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 20 (Actual)
Dates: Start 2010-01; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
static balance | after one session, four and eight weeks

SECONDARY OUTCOMES:
reaction time | after one session, after four and eight weeks
dynamic balance | after one session, four and eight weeks

REFERENCES:
- [Result] Rogan S, Hilfiker R, Schmid S, Radlinger L. Stochastic resonance whole-body vibration training for chair rising performance on untrained elderly: a pilot study. Arch Gerontol Geriatr. 2012 Sep-Oct;55(2):468-73. doi: 10.1016/j.archger.2012.02.011. Epub 2012 Mar 16. PMID 22425243
- [Result] Rogan S, Radlinger L, Schmid S, Herren K, Hilfiker R & de Bruin ED. Skilling up for training: a feasibility study investigating acute effects of stochastic resonance whole-body vibration on postural control of older adults. Ageing Research. 2012;3(1):e5
- [Derived] Rogan S, Radlinger L, Hilfiker R, Schmidtbleicher D, de Bie RA, de Bruin ED. Feasibility and effects of applying stochastic resonance whole-body vibration on untrained elderly: a randomized crossover pilot study. BMC Geriatr. 2015 Mar 12;15:25. doi: 10.1186/s12877-015-0021-4. PMID 25886789